CLINICAL TRIAL: NCT00477893
Title: Can New Imaging- and Bio-markers Improve the Assessment of Disease Activity and Progression and Predict Therapeutic Outcome in Spondyloarthritis Patients Receiving Adalimumab
Brief Title: Danish Multicenter Study of Adalimumab in Spondyloarthritis
Acronym: DANISH
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, MOstergaard, Professor, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUM 04-078
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Adalimumab (Active Comparator)
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — sc. injection Humira 40 mg every other week, from week 0 or 12 to the end of study
  Arms: Adalimumab
Drug: Placebo — sc. inj. placebo every other week, week 0, 2, 4, 6, 8, and 10.
  Arms: Placebo

SUMMARY:
Spondyloarthropathies (SpA) are often diagnosed with a considerable delay (often 8-10 years from symptom onset), because the available clinical, biochemical and radiological methods are not sufficiently sensitive. TNF-a antagonists have recently been introduced for treatment of SpA, and current data indicate a higher efficacy than previously available therapies. The improved treatment options have increased the need for improved methods for diagnosis, monitoring and prognostication of these diseases, so that the efficient therapies can be initiated at the optimal time point and monitored optimally. Magnetic resonance imaging (MRI) and a number of biomarkers are promising, but not yet sufficiently studied, methods for this.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of spondyloarthritis according to the European Spondyloarthritis Study Group (ESSG) criteria
2. Clinical active disease, defined as a BASDAI score > 4 despite concurrent NSAID therapy
3. Presence of sacroiliitis on conventional radiography or MRI.
4. Among other issues: Age >18 years; adequate birth control; no contraindications for anti-TNFa-therapy, no previous TNFa-antagonists

Exclusion Criteria:

1. Previous TNFα inhibitor therapy
2. Treatment with disease modifying anti-rheumatic drugs within 4 weeks before screening
3. Oral, intraarticular, intramuscular or intravenous glucocorticoid within 4 weeks before screening
4. Pregnancy or lactation
5. HIV, hepatitis B or C, tuberculosis, other infections
6. Malignancies
7. Other serious concomitant diseases (uncontrolled/severe kidney, liver, haematological, gastrointestinal, endocrine, cardiovascular, pulmonary, neurological ore cerebral disease (including demyelinating disease)
8. Contraindications to anti-TNFa-therapy
9. Contraindications to MRI

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in BASDAI of 20 mm or 50% | 12-24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Inge Juul Sørensen, Dr., Study Chair — Department of Rheumatology, Glostrup University Hospital; Susanne Juhl Pedersen, Dr., Study Chair — Department of Rheumatology, Glostrup University Hospital; Mikkel Ostergaard, Professor, Principal Investigator — Department of Rheumatology, Glostrup University Hospital
Locations (13):
- Denmark (13):
  - Department of Radiology, Aabenraa Hospital, Aabenraa
  - Department of Radiology, Århus University Hospital, Aarhus
  - Department of Radiology, Herlev University Hospital, Copenhagen
  - Department of Rheumatology, Bispebjerg University Hospital, Copenhagen
  - Department of Rheumatology, Gentofte University Hospital, Copenhagen
  - Department of Rheumatology, Glostrup University Hospital, Copenhagen
  - Department of Rheumatology, Herlev University Hospital, Copenhagen
  - Department of Rheumatology, Hvidovre University Hospital, Copenhagen
  - King Christian X´s Hospital of Rheumatic Diseases, Gråsten
  - Department of Rheumatology, Hørsholm Hospital, Hørsholm
  - Department of Rheumatology, Slagelse Hospital, Slagelse
  - Department of Radiology, Vejle Hospital,, Vejle
  - Department of Rheumatology, Vejle Hospital, Vejle

REFERENCES:
- [Derived] Pedersen SJ, Poddubnyy D, Sorensen IJ, Loft AG, Hindrup JS, Thamsborg G, Asmussen K, Hendricks O, Norregaard J, Piil AD, Moller JM, Jurik AG, Balding L, Lambert RG, Sieper J, Ostergaard M. Course of Magnetic Resonance Imaging-Detected Inflammation and Structural Lesions in the Sacroiliac Joints of Patients in the Randomized, Double-Blind, Placebo-Controlled Danish Multicenter Study of Adalimumab in Spondyloarthritis, as Assessed by the Berlin and Spondyloarthritis Research Consortium of Canada Methods. Arthritis Rheumatol. 2016 Feb;68(2):418-29. doi: 10.1002/art.39434. PMID 26414004